CLINICAL TRIAL: NCT03179657
Title: Guangzhou Nutrition and Health Study (GNHS): A Multiomics-based Study
Brief Title: Guangzhou Nutrition and Health Study (GNHS)
Acronym: GNHS
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yu-ming Chen, Professor, Sun Yat-sen University
Other Study IDs: 2007032
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Cardiovascular Diseases; Osteoporosis; Diabetes Mellitus, Type 2; Metabolic Syndrome; Obesity; Hypertension; Non-Alcoholic Fatty Liver Disease; Chronic Kidney Diseases; Cancer; Death; Nutrition Disorders; Sarcopenia
Keywords: Prospective Cohort study; Nutrition; Diet; Multi-omics; Metabolic diseases; Guangzhou; Chinese
MeSH Terms: conditions — Cardiovascular Diseases; Osteoporosis; Diabetes Mellitus, Type 2; Metabolic Syndrome; Obesity; Hypertension; Non-alcoholic Fatty Liver Disease; Renal Insufficiency, Chronic; Neoplasms; Death; Nutrition Disorders; Sarcopenia; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 12-h fasting venous blood, urine, feces and saliva were/will be collected at baseline and follow-ups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: The Guangzhou Nutrition and Health Study (GNHS) project aims to assess the determinants of metabolic disease in nutritional aspects, as well as other environmental and genetic factors, and explore possible mechanisms with multi-omics integration.

Study design: GNHS is a community-based prospective cohort study. Participants: In this cohort, the original GNHS and another cohort study (the controls of a case-control study of hip fractures, CCFH) have been integrated into the one GNHS project. After completing the baseline examination, a total of 5118 participants were recruited during 2008-2015 in the GNHS project.

Visits and Data Collection: Participants were/will be visited every three years by invited to the School of Public Health, Sun Yat-sen University. At each visit, face-to-face interviews, specimen collection, anthropometric measurements, dual-energy x-ray absorptiometry (DXA) scanning, ultrasonography evaluation, vascular endothelial function evaluation, cardiopulmonary exercise testing, magnetic resonance imaging (MRI), 14-d real-time continuous glucose monitoring tests, laboratory tests, and multi-omics data were/will be conducted. Up to December 2022, 3442 and 2895 subjects completed the 2nd and 3rd visits.

Key variables:

1. Questionnaire interviews.
2. Physical examinations: Anthropometric measurements, blood pressure tests, handgrip strength, muscle function and bracelet motion monitoring.
3. DXA scanning: To determine bone density, bone mineral content, bone geometry information, fat mass, and muscle mass.
4. Ultrasonography evaluations: To determine carotid artery intima-media thickness and plaque, and fatty liver.
5. Vascular endothelial function evaluation.
6. Cardiopulmonary exercise testing: Lung function.
7. MRI: Brain and upper-abdomen MRI.
8. 14-d Real-time continuous glucose monitoring tests.
9. Specimen collections: Overnight fasting blood, early morning first-void urine, faces, and saliva samples.
10. Laboratory tests: Metabolic syndrome-related indices; Diabetes-related indices; Uric acid; Nutritional indices; Inflammatory cytokines; Index of oxidative stress; Adipocytes; Sexual hormones; Liver and renal function-related markers; Routine blood test.
11. Multi-omics data: Genotyping data; Gut microbiota; Untargeted serum and fecal proteomics; Targeted serum and fecal metabolomics.
12. Morbidity and mortality: Relevant data were/will be also retrieved via local multiple health information systems.

DETAILED DESCRIPTION:
Purpose: The Guangzhou Nutrition and Health Study (GNHS) aims to assess the determinants of risk of metabolic diseases and changes in their relevant indices (e.g., osteoporosis, atherosclerosis, type 2 diabetes, hypertension, metabolic syndrome, non-alcoholic fatty liver disease, cardiovascular diseases, chronic kidney disease, body composition, lung function, cognition function, etc.) in nutritional aspects, as well as other environmental and genetic factors.

Study design: GNHS is a community-based prospective cohort study. Participants: In this cohort, the original GNHS and another cohort study (the controls of a case-control study of hip fractures, CCFH) have been integrated into the one GNHS project. About 4048 apparently healthy residents (aged 40-80 years) in the original GNHS were recruited between 2008 and 2013, and 1070 participants in the CCFH baseline (52-83 years old) were recruited from 2009 to 2015, all living in Guangzhou city (South China) for >5 years. After completing the baseline examination, a total of 5118 participants were recruited during 2008-2015 in the GNHS project.

Visits and Data Collection: Participants were/will be visited every three years by invited to the School of Public Health, Sun Yat-sen University. At each visit, face-to-face interviews, specimen collection, anthropometric measurements, DXA scanning, ultrasonography evaluation, vascular endothelial function evaluation, cardiopulmonary exercise testing, MRI, 14-d real-time continuous glucose monitoring tests, laboratory tests, and multi-omics data were/will be conducted. Up to December 2022, 3442 and 2895 subjects completed the 2nd and 3rd visits. The 4th visit began in 2017 and has been ongoing, and 2243 participants have been revisited so far. About 1500 participants responded in 2020-now at the 5th visit. It is planned to follow up the participant in person for at least 15 years.

Key variables:

1. Questionnaire interviews: Structured questionnaires were/will be used to collect the participants' socio-demographic characteristics (e.g., age, sex and household income), lifestyle factors (smoking, passive smoking, alcohol drinking, tea drinking, physical activity), menstruation and reproductive history (women only), sleep quality (Pittsburgh Sleep Quality Index, PSQI), family history, psychological health (Self-Rating Anxiety Scale, SAS), Simplified Geriatric Depression Scale (GDS), social support and participation, cognitive function (Mini-Mental State Examinations (MMSE), and Addenbrooke's cognitive examination (ACE)), habitual dietary intake (a validated 79-item quantitative food frequency questionnaire), use of supplements and history of chronic diseases.
2. Physical examinations: Anthropometric measurements (weight, height, waist, hip and neck circumference, etc.), blood pressure tests, handgrip strength, muscle function and bracelet motion monitoring.
3. DXA scanning: A dual-energy x-ray absorptiometry (DXA, Discovery W; Hologic Inc.) was/will be used to determine bone density and bone mineral content at the whole body, lumbar spine (L1-L4), left hip sites, bone geometry information at the hip, fat mass and muscle mass at total body and its sub-regions.
4. Ultrasonography evaluations: Ultrasonography evaluation of the carotid artery and upper abdominal organs (e.g., liver and kidney) was/will be performed to determine carotid artery intima-media thickness and plaque, fatty liver.
5. Vascular endothelial function evaluation: Blood flow-mediated vasodilation.
6. Cardiopulmonary exercise testing: Lung function.
7. MRI: Magnetic resonance imaging in the brain was/will be used to study brain tissue's microstructure and investigate brain function. Upper-abdomen MRI was/will be conducted to assess the structure and contents of fat and iron of the liver, fat and muscle mass, and vertebral bone marrow fat, and help to identify renal angiomyolipoma and malignant renal tumours.
8. 14-d Real-time continuous glucose monitoring tests: A 14-d continuous glucose monitoring was used to determine glycemic responses to various usual daily foods (by a 7-d image-based food diary) using 3-type standard breakfast as internal calibrators.
9. Specimen collections: Overnight fasting blood sample was/will be collected and separated into serum, plasma, erythrocyte and leukocyte within two hours. Early morning first-void urine, faces, and saliva samples were/will be collected, separated and stored at -80°C till tests.
10. Laboratory tests:

    1. Fasting serum lipid profile.
    2. Diabetes-related indices; fasting glucose, insulin, HbA1c, and fructosamine.
    3. Uric acid.
    4. Nutritional indices: fatty acids, vitamins, minerals, alkaloids, carotenoids, flavonoids, sulfur-containing amino acids and so on.
    5. Inflammatory cytokines.
    6. Index of oxidative stress.
    7. Adipocytes.
    8. Sexual hormones.
    9. Liver and renal function-related markers.
    10. Routine blood test.
11. Multi-omics data:

    1. Genotyping data (Illumina Asian Screening-750000 arrays).
    2. Gut microbiota: 16S ribosomal RNA, metagenome, and internal transcribed spacer 2 (ITS2) sequencing.
    3. Untargeted serum and fecal proteomics: about 430 unique human protein groups in serum, 1253 human protein and 83683 microbial proteins in feces.
    4. Targeted serum and fecal metabolomics: amino acids, benzenoid, bile acids, carbohydrates, carnitines, fatty acids, indoles, nucleosides, organic acids, organooxygen compounds, phenylpropanoic acids, pyridines and so on. Approximately 200 metabolites have been quantified so far.
12. Morbidity and mortality: Relevant data were/will be also retrieved via local multiple health information systems.
13. Others: Many other laboratory tests or instrument tests will be developed depending on needs and resources in future.

Data analysis: Analyses of variance and covariance, or mixed effects model were/will be used to compare the mean differences in continuous outcomes (e.g., changes of bone mineral density, body fat mass, or intima-media thickness) among the quartiles. Cox proportional hazards or logistic regression models were/will be used to assess the risk of exposures (e.g., nutrition intakes and physical activity) on categorical outcomes. Path analysis was/will be used to assess the potential mediating effects in the causal pathway between exposures and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-80 years (the original GNHS) and 40-85 years (CCFH) at baseline;
* Living in Guangzhou for at least five years;
* Chinese.

Exclusion Criteria:

* Had a history of hospital-confirmed diabetes, failure(s) of heart, liver, or kidney, cancer, cardiovascular events, metabolic bone diseases, glucocorticoid use (over 3 mo.) or sexual hormone use (over 6 mo.), spine or hip fractures;

On special diet due to a disease or weight control;

* Mental and physical disability;
* Likely to move to other city within 5 years;
* Did not want to attend any one item of the survey or sample collection.

Ages: 40 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 4048 participants in the original GNHS (79.1%) and 1070 participants in the CCFH (20.9%) contributed to the GNHS project (5118 participants). The sample of the GNHS project consisted of 68.1% women. At baseline, the median age was 59.0 years. 41.6% and 23.4% of them had education levels of secondary high school and college degree or above. 86.2% were married and 15.8% were smokers. Median BMI was 23.2 kg/m2. Up to December 2022, 5118 participants attended baseline survey, 3442 and 2895 subjects completed the 2nd and 3rd visits. The whole cohort is planned to be followed at least 15 years.
Sampling Method: Non-Probability Sample
Enrollment: 5118 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular diseases (change in carotid artery intima-media thickness, and occurrence of cardiovascular diseases) | Up to 15 years
  The investigators will track for occurrence of cardiovascular diseases by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Guangzhou Center for Disease Control and Prevention, and Health Insurance Bureau. All cases will be verified by medical record reviews. The investigators will also measure the carotid artery intima-media thickness at each visit (every 3 years)，and analyze the change of carotid artery intima-media thickness.
Bone health (change of bone mineral density, and occurrence of osteoporosis and fractures) | Up to 12 years
  The investigators will measure the bone mineral density at each follow-up, and osteoporosis was defined as T-score ≤ -2.5 in accordance with the World Health Organization criteria. The investigators will also track for occurrence of osteoporosis and fractures by follow-up surveys and annual record linkage to the population-based disease or death registration collected by the Guangzhou Center for Disease Control and Prevention, and Health Insurance Bureau. All cases will be verified by medical record reviews. Moreover, the investigators will analysis the annual change of bone mineral density.
Nonalcoholic fatty liver disease (NAFLD) | Up to 12 years
  The investigators will measure the abdominal ultrasonography at each follow-up and NAFLD was diagnosed based on standard criteria issued by the Fatty Liver Disease Study Group of the Chinese Liver Disease Association. The upper-abdomen MRI was conducted in the 5th visit and NAFLD was diagnosed based on proton density fat fraction. The investigators will also track for occurrence of NAFLD by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Guangzhou Center for Disease Control and Prevention and Health Insurance Bureau. All cases will be verified by medical record reviews.

SECONDARY OUTCOMES:
Change in adiposity-related indices | Up to 12 years
  The investigators will measure the anthropometric indices at each visit and DXA-derived body fat composition since the 2nd visit. And the investigators will also analyze the change of adiposity-related indices.
Metabolic syndrome | Up to 15 years
  The investigators will measure metabolic syndrome-related indices at each visit (every 3 years), and the investigators can analyze the incidence of metabolic syndrome and the changes of the individual items.
Change in muscle mass | Up to 12 years
  The investigators will measure the DXA-derived body muscle since Visit 2. And the investigators will also analyze the change of adiposity-related indices.
Sarcopenia | Up to 12 years
  The investigators will measure the handgrip strength, usual gait speed, and DXA-derived body muscle since Visit 2. The sarcopenia will be diagnosed according to definition recommended by Asian Working Group for Sarcopenia (AWGS): cutoff values for muscle mass measurements (7.0 kg/m2 for men and 5.4 kg/m2 for women by using dual X-ray absorptiometry, and 7.0 kg/m2 for men and 5.7 kg/m2 for women by using bioimpedance analysis), handgrip strength (<26 kg for men and <18 kg for women), and usual gait speed (<0.8 m/s).
Diabetes mellitus (change of diabetic indices) | Up to 15 years
  The investigators will measure the blood glucose, insulin, and HbA1C. The investigators will also track for occurrence of diabetes mellitus by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Guangzhou Center for Disease Control and Prevention and Health Insurance Bureau. All cases will be verified by medical record reviews. Moreover, the investigators also will analyze the annual change of blood glucose and other diabetic indices.
Cancer | Up to 15 years
  The investigators will track for cancer occurrence by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Guangzhou Center for Disease Control and Prevention and Health Insurance Bureau. All cases will be verified by medical record reviews.
Chronic kidney disease (CKD) | Up to 12 years
  The investigators will measure the serum creatine and urine creatine and protein at baseline and each follow-up and CKD will be defined as an estimated glomerular filtration rate of <60 mL/min/1.73 m2 or and the presence of an elevated urine microalbumin/creatinine ratio. The investigators will also track for occurrence of CKD by follow-up surveys and annual record linkage to the population-based disease or death registry collected by the Guangzhou Center for Disease Control and Prevention and Health Insurance Bureau. All cases will be verified by medical record review.
Cognitive function | Up to 6 years
  The investigators will measure the cognitive function using questionnaires (Mini-Mental State Examinations / Addenbrooke's cognitive examination) at the 4th and 5th visits and brain MRI at the 5th visit. The investigators will also track for annual record linkage to the population-based disease or death registry collected by the Guangzhou Center for Disease Control and Prevention and Health Insurance Bureau.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Chen, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Z, Huang BX, Huang ZH, Li MC, Chen YM, Zhu HL. Exploring the link between serum betaine levels and hyperuricemia risk in middle-aged and older adults: insights from a prospective cohort study. Eur J Nutr. 2025 Feb 1;64(2):77. doi: 10.1007/s00394-025-03594-0. PMID 39891737
- [Derived] Xie K, Xiao C, Lin L, Li F, Hu W, Yang Y, Chen D, Miao Z, Sun TY, Yan Y, Zheng JS, Chen YM. Erythrocyte Very Long-Chain Saturated Fatty Acids, Gut Microbiota-Bile Acid Axis, and Incident Coronary Artery Disease in Adults: A Prospective Cohort Study. J Nutr. 2024 Oct;154(10):3019-3030. doi: 10.1016/j.tjnut.2024.08.005. Epub 2024 Aug 10. PMID 39128547
- [Derived] Chen S, Chen XY, Huang ZH, Fang AP, Li SY, Huang RZ, Chen YM, Huang BX, Zhu HL. Correlation between serum trimethylamine-N-oxide and body fat distribution in middle-aged and older adults: a prospective cohort study. Nutr J. 2024 Jul 9;23(1):70. doi: 10.1186/s12937-024-00974-w. PMID 38982486
- [Derived] Chen S, Lin X, Ma J, Li M, Chen Y, Fang AP, Zhu HL. Dietary protein intake and changes in muscle mass measurements in community-dwelling middle-aged and older adults: A prospective cohort study. Clin Nutr. 2023 Dec;42(12):2503-2511. doi: 10.1016/j.clnu.2023.10.017. Epub 2023 Oct 22. PMID 37922694
- [Derived] Wu YY, Gou W, Yan Y, Liu CY, Yang Y, Chen D, Xie K, Jiang Z, Fu Y, Zhu HL, Zheng JS, Chen YM. Gut microbiota and acylcarnitine metabolites connect the beneficial association between equol and adiposity in adults: a prospective cohort study. Am J Clin Nutr. 2022 Dec 19;116(6):1831-1841. doi: 10.1093/ajcn/nqac252. PMID 36095141
- [Derived] Li SY, Chen S, Lu XT, Fang AP, Chen YM, Huang RZ, Lin XL, Huang ZH, Ma JF, Huang BX, Zhu HL. Serum trimethylamine-N-oxide is associated with incident type 2 diabetes in middle-aged and older adults: a prospective cohort study. J Transl Med. 2022 Aug 18;20(1):374. doi: 10.1186/s12967-022-03581-7. PMID 35982495
- [Derived] Gu Y, Luo J, Chen Q, Qiu Y, Zhou Y, Wang X, Qian X, Liu Y, Xie J, Xu Z, Ling W, Chen Y, Yang L. Inverse Association of Serum Adipsin with the Remission of Nonalcoholic Fatty-Liver Disease: A 3-Year Community-Based Cohort Study. Ann Nutr Metab. 2022;78(1):21-32. doi: 10.1159/000520368. Epub 2021 Nov 23. PMID 34814152
- [Derived] Deng YY, Zhong QW, Zhong HL, Xiong F, Ke YB, Chen YM. Higher Healthy Lifestyle Score is associated with lower presence of non-alcoholic fatty liver disease in middle-aged and older Chinese adults: a community-based cross-sectional study. Public Health Nutr. 2021 Oct;24(15):5081-5089. doi: 10.1017/S1368980021000902. Epub 2021 Feb 26. PMID 33634772
- [Derived] Xiao ML, Lin JS, Li YH, Liu M, Deng YY, Wang CY, Chen YM. Adherence to the Dietary Approaches to Stop Hypertension (DASH) diet is associated with lower presence of non-alcoholic fatty liver disease in middle-aged and elderly adults. Public Health Nutr. 2020 Mar;23(4):674-682. doi: 10.1017/S1368980019002568. Epub 2019 Sep 30. PMID 31566148
- [Derived] Dong HL, Tang XY, Deng YY, Zhong QW, Wang C, Zhang ZQ, Chen YM. Urinary equol, but not daidzein and genistein, was inversely associated with the risk of type 2 diabetes in Chinese adults. Eur J Nutr. 2020 Mar;59(2):719-728. doi: 10.1007/s00394-019-01939-0. Epub 2019 Apr 5. PMID 30953148
- [Derived] Chen ZY, Liu M, Jing LP, Xiao ML, Dong HL, Chen GD, Chen YM. Erythrocyte membrane n-3 polyunsaturated fatty acids are inversely associated with the presence and progression of nonalcoholic fatty liver disease in Chinese adults: a prospective study. Eur J Nutr. 2020 Apr;59(3):941-951. doi: 10.1007/s00394-019-01953-2. Epub 2019 Apr 1. PMID 30937580
- [Derived] Xiao ML, Chen GD, Zeng FF, Qiu R, Shi WQ, Lin JS, Cao Y, Li HB, Ling WH, Chen YM. Higher serum carotenoids associated with improvement of non-alcoholic fatty liver disease in adults: a prospective study. Eur J Nutr. 2019 Mar;58(2):721-730. doi: 10.1007/s00394-018-1678-1. Epub 2018 Mar 29. PMID 29594435